CLINICAL TRIAL: NCT06854549
Title: The Effectiveness of Parental Reading Picture-book Intervention on Cardiopulmonary Stability, Hospitalization Anxiety and Parent-Child Attachment Relationship With Premature Infants
Brief Title: Impact of Picture Book Reading on Preterm Infant Stability, Parental Anxiety, and Parent-Child Attachment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-02-002A
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-06

CONDITIONS: Effects of Parent-Child Reading on Preterm Infant Stability, Parental Anxiety, and Parent-Child Attachment
Keywords: Reading Picture-book; Premature Infants; Hospitalization anxiety; Cardiopulmonary stability; parent-child attachment relationship
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preterm Infant Stability, Parental Anxiety, Parent-Child Attachment (Experimental)
  Interventions: Behavioral: Parental Reading Picture-book
- Routine Care (No Intervention): The control group in this study will receive standard routine care in the neonatal ward and intensive care unit of a medical center in Northern Taiwan. Routine clinical care involves one parent visiting the preterm infant during visiting hours. After the physician or nurse explains the infant's current condition to the parent, the parent is allowed to visit the preterm infant freely for half an hour. On the day of discharge, control group participants will receive the same educational booklet titled "Reading Picture Books from Scratch" as the experimental group. The benefits and importance of picture book reading interventions will be explained to them, and parents will be encouraged to use the gifted picture books for reading activities at home.

INTERVENTIONS:
Behavioral: Parental Reading Picture-book — In addition to receiving routine care, the experimental group will be given the "Reading Picture Books from Scratch" educational booklet once the preterm infant is removed from the incubator, the group assignment is confirmed, and participation in the study is verified. They will then undergo the "Picture Book Reading Intervention." This intervention targets the preterm infant and one of the parents. It involves reading picture books from the second to the fourth day after the infant is removed from the incubator, during the visiting period from 14:10 to 14:20.
  Other Names: Experimental Group
  Arms: Preterm Infant Stability, Parental Anxiety, Parent-Child Attachment

SUMMARY:
This study investigates the effects of a parent-child picture book reading intervention on the cardiopulmonary stability of preterm infants, parental anxiety, and parent-child attachment. A randomized controlled trial will be conducted in a neonatal intensive care unit (NICU) and neonatal intermediate care unit in northern Taiwan. A total of 88 preterm infants and their parents will be randomly assigned to an intervention or control group. Parents in the intervention group will read picture books to their infants from a corrected gestational age of 28 weeks to 36 weeks and 6 days. Physiological data (heart rate, respiratory rate, oxygen saturation, and heart rate variability) and parental anxiety levels will be assessed at multiple time points. The study aims to determine whether this intervention improves infant stability, reduces parental anxiety, and enhances parent-child attachment, contributing to improved neonatal care practices.

DETAILED DESCRIPTION:
Background The birth and survival rates of preterm infants in our country have significantly improved. However, due to the immaturity of their autonomic nervous systems, preterm infants are at risk of complications stemming from unstable vital signs. This instability often induces anxiety in parents, which can further impact their psychological adjustment and hinder the establishment of a secure parent-child attachment. Consequently, this study aims to develop a systematic intervention program using picture book reading to improve the cardiopulmonary stability of preterm infants, alleviate parental anxiety, and enhance the parent-child bond.

Objective To evaluate the effects of a parent-child picture book reading intervention on the cardiopulmonary stability of preterm infants, parental anxiety during hospitalization, and the parent-child attachment relationship.

Methods This study will employ a randomized controlled trial (RCT) design. Participants will include preterm infants and at least one parent from the neonatal intensive care unit (NICU) and neonatal intermediate care unit of a medical center in northern Taiwan. A total of 88 pairs of preterm infants and their parents will be recruited and randomly assigned to either the experimental or control group. The intervention consists of parents reading picture books to their preterm infants, starting at a corrected gestational age of 28 weeks and continuing until 36 weeks and 6 days. Data will be collected at multiple time points, including measurements of heart rate, respiratory rate, oxygen saturation, and heart rate variability. Subjective data will be gathered using the State-Trait Anxiety Inventory (STAI) and the Parent-Child Attachment Scale, while objective data will be recorded via physiological monitors and heart rate variability analyzers. Statistical analyses, including independent samples t-tests, repeated measures ANOVA, and generalized estimating equations (GEE), will be performed to compare the intervention's effectiveness.

Project Goal To develop and evaluate the effectiveness of a parent-child picture book reading intervention program for preterm infants. The findings aim to inform pediatric clinical care practices and support the health and well-being of families with preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm Infants:

  1. Born between 28+0 and 36+6 weeks of gestation.
  2. Transferred out of the incubator as per medical advice.
  3. Passed the newborn hearing screening in both ears.
* Parents of Preterm Infants:

  1. Able to read and comprehend Chinese-language materials.
  2. Capable of communicating in Mandarin.

Exclusion Criteria:

* Preterm Infants:

  1. Presence of external ear abnormalities.
  2. Receiving sedatives, hypnotics, or caffeine therapy.
* Parents of Preterm Infants:

  1. Having auditory or speech impairments.

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary stability | ecorded at 14:00, 14:10, and 14:20 on the second to fourth days after incubator transfer, as well as at 14:20 on the fifth day.
  The intervention period in this study begins on the second day after the preterm infant is transferred out of the incubator and concludes on the fifth day. Data collection occurs at 24 time points throughout the study. Physiological indicators, including heart rate, respiratory rate, oxygen saturation, and heart rate variability, are recorded at 14:00, 14:10, and 14:20 on the second to fourth days after incubator transfer, as well as at 14:20 on the fifth day.

SECONDARY OUTCOMES:
Hospitalization anxiety | After confirming the assigned group, and research Day 5
  After group assignment is confirmed, the parents of the participants complete the pretest questionnaire of the State-Trait Anxiety Inventory (STAI). On the fifth day of the study, they complete the posttest questionnaire of the State Anxiety Scale.
  The STAI consists of 20 items, scored using a 4-point Likert scale: 1 ("Not at all"), 2 ("Somewhat"), 3 ("Moderately so"), and 4 ("Very much so"). The total score is the sum of all item scores, with higher scores indicating higher levels of anxiety. A total score of 20-39 indicates mild anxiety, 40-59 indicates moderate anxiety, and 60 or above indicates severe anxiety.
parent-to-infant attachment | After group assignment is confirmed ,and the fifth day of the study.
  After group assignment is confirmed, the parents of the participants complete the pretest questionnaire of the "Maternal Attachment Inventory". On the fifth day of the study, they complete the posttest questionnaire of the "Maternal Attachment Inventory(MAI)".
  The MAI consists of 22 items, scored using a 4-point scale ranging from 1 ("Almost never") to 4 ("Almost always"). The total score ranges from 22 to 88, with higher scores indicating a stronger mother-infant attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Jy Jeng, PhD, Study Chair — Taipei Veterans General Hospital, Taipei
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou, Taiwan

IPD SHARING:
Plan to Share IPD: No